CLINICAL TRIAL: NCT06926192
Title: Efficacy and Safety of Secukinumab in Conjunction With Surgery in Moderate to Severe Hidradenitis Suppurativa: An Open-label Cohort Study in Real Clinical Practice
Brief Title: Efficacy and Safety of Secukinumab in Conjunction With Surgery in Moderate to Severe Hidradenitis Suppurativa
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Junyou ZHENG, Dr, Peking Union Medical College
Other Study IDs: 2025-KY-016
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Hidradenitis Suppurativa (HS); Hidradenitis Suppurativa (Acne Inversa); Secukinumab
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — secukinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Moderate to severe hidradenitis suppurativa
  Interventions: Combination Product: Surgery combined with secukinumab

INTERVENTIONS:
Combination Product: Surgery combined with secukinumab — Surgery combined with secukinumab

SUMMARY:
This study aims to retrospectively analyze the efficacy and safety of secukinumab combined with surgery in treating moderate to severe HS in real-world clinical practice, providing clinical practioners with real-world evidence in HS treatment.

DETAILED DESCRIPTION:
Hidradenitis suppurativa (HS) is a chronic, recurrent, and disabling inflammatory disease that occurs in apocrine distribution sites such as the axilla, groin, and perianal region with a worldwide prevalence of approximately 1.5% -4.6%.The pathogenesis is excessive activation of the Th17 type immune response mediated by IL-17, IL-23, resulting in abnormal keratinization of hair follicles, obstruction of sebaceous ducts, and bacterial infection, culminating in abscesses, sinus tracts, and scarring.Patients with moderate to severe HS (Hurley stage II-III) often suffer from a severe decline in their quality of life due to recurrent infections, pain, and dysfunction, and their risk of depression is markedly elevated.Traditional treatments such as antibiotics, glucocorticoids, surgical debridement have limited efficacy, and the recurrence rate of surgery alone is as high as 50% -70%.In recent years, the use of biologic agents such as TNF-α inhibitors has dramatically improved HS outcomes, but 30% to 40% of patients still have an inadequate response to TNF-α inhibitors. Accumulating evidence suggests that the IL-17 pathway plays a key role in HS pathogenesis, that IL-17A expression is upregulated in the skin lesions of HS patients and positively correlates with disease severity. The efficacy and safety of secukinumab in combination with surgery remain unclear.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 80 years old with moderate-severe (Hurley II-III) HS
2. The diagnosis of HS was confirmed by histopathological examination in the Department of Pathology of our hospital
3. Patients with HS who received secukinumab combined with surgery in the Department of Dermatologic Surgery of our hospital
4. Patients with complete clinical data followed up for at least 1 year

Exclusion Criteria:

1. Patients lost to follow-up
2. Patients with less than one year of follow-up
3. Patients who received additional adjuvant therapy during the follow-up period

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged 18 to 80 years old with moderate-severe (Hurley II-III) HS
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-06-21 (Estimated)

PRIMARY OUTCOMES:
HiSCR | week 52
  at least a 50% reduction in total AN count, with no increase in abscess count, and no increase in draining fistula count relative to baseline)

SECONDARY OUTCOMES:
IHS4 | week 52
  the number of nodules (multiplied by 1) plus the number of abscesses (multiplied by 2) plus the number of draining tunnels (multiplied by 4)
Change in number of inflammatory nodules | week 52
  Change in number of inflammatory nodules
Change in number of abscesses | week 52
  Change in number of abscesses
Change in number of sinus tracts | week 52
  Change in number of sinus tracts
HS related skin pain (NRS30) | week 52
  NRS30 is defined as at least a 30% reduction from baseline and at least a 2-unit reduction in patient's global assessment of skin pain at worst
Time to onset of action | week 52
  Time to onset of action
Duration of drug effect | week 52
  Duration of drug effect
Changes in inflammatory markers | week 52
  white blood cells, erythrocyte sedimentation rate, C-reactive protein
DLQI | week 52
  Dermatology Life Quality Index
WPAI | week 52
  Work Productivity and Activity Impairment
Adverse effect and complications | week 52
  Adverse effect and complications

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Skin Diseases, Institute of Dermatology, Chinese Academy of Medical Science and Peking Union Medical College, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fang V, Gupta R, Micheletti RG. Managing Hidradenitis Suppurativa with Biologics and Small Molecule Inhibitors. Dermatol Clin. 2025 Apr;43(2):231-245. doi: 10.1016/j.det.2024.12.008. Epub 2025 Jan 21. PMID 40023624
- [Background] Calabrese L, Cartocci A, Rubegni P, French LE, Kendziora B. Efficacy and safety of biologics for hidradenitis suppurativa: A network meta-analysis of phase III trials. J Eur Acad Dermatol Venereol. 2025 Mar 10. doi: 10.1111/jdv.20617. Online ahead of print. PMID 40062409
- [Background] Kohorst JJ, Baum CL, Otley CC, Roenigk RK, Pemberton JH, Dozois EJ, Tran NV, Davis MD. Patient Satisfaction and Quality of Life Following Surgery for Hidradenitis Suppurativa. Dermatol Surg. 2017 Jan;43(1):125-133. doi: 10.1097/DSS.0000000000000942. PMID 28027202
- [Background] Caliezi A, Rabufetti A, Hunger R, Wolf R, Seyed Jafari SM. Impact of Hidradenitis Suppurativa on Sexual Quality of Life. J Clin Med. 2025 Jan 30;14(3):910. doi: 10.3390/jcm14030910. PMID 39941581
- [Background] Agnese ER, Tariche N, Sharma A, Gulati R. The Pathogenesis and Treatment of Hidradenitis Suppurativa. Cureus. 2023 Nov 25;15(11):e49390. doi: 10.7759/cureus.49390. eCollection 2023 Nov. PMID 38146560
- [Background] Jemec GB. Clinical practice. Hidradenitis suppurativa. N Engl J Med. 2012 Jan 12;366(2):158-64. doi: 10.1056/NEJMcp1014163. No abstract available. PMID 22236226